CLINICAL TRIAL: NCT03842852
Title: Comparition of the Results of Inguinal Hernia Repair Using Laparoscopic Total Extra-peritoneal or Open Prolene Hernia System Approach
Brief Title: Laparoscopic TEP (Total Extra-peritoneal) Repair Vs Open PHS (Prolene Hernia System)
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the department of general surgery, Assuta Medical Center
Other Study IDs: 02-19
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; laparoscopy reapir; open repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LTEPR: Patients who underwent inguinal hernia repair laparoscopic extra-peritoneal repair under general anesthesia.
  Interventions: Procedure: Inguinal hernia repair
- OPHSR: Patients that underwent inguinal hernia repair open using prolene hernia system mesh under general or regional anesthesia.
  Interventions: Procedure: Inguinal hernia repair

INTERVENTIONS:
Procedure: Inguinal hernia repair — The grupo one underwent open repair and laparoscopic repair

SUMMARY:
Abdominal wall hernias are common, with a lifetime risk of 27% in men and 3% in women.

Inguinal and femoral hernias are the most common affections faced by primary care physicians that require surgical intervention.

The most common hernia in both sexes is the indirect inguinal hernia. The male-to-female ratio is 9:1 for inguinal hernias and 1:3 for femoral hernias. Inguinal hernia repair is one of the most common operations undertaken in routine surgical practice.

Since the introduction of the Bassini method in 1887, more than 70 types of pure tissue repair have been reported in the surgical literature. Throughout the years, attention was paid to the recurrences that occur after the use of tissue approximation technique, in the literature it has been reported that they occur in up to 34% of cases, being that the actual incidence of recurrences it is underreported, therefore, the repair of the hernia with approximation of tissue has practically been abandoned.

The concept of tension free repair for hernias was introduced by Lichtenstein who explain that the prime etiologic factor behind most herniorrhaphy failures is the suturing together, under tension, of structures that are not normally in apposition. The technique of the hernioplasty with the use of mesh was not widely accepted at first, the expansion of the use of mesh expanded for years. The use of mesh increased from 7 per cent of all operations in 1992 to 51 per cent in 1996. Currently, groin hernia treatment is not standardized but, today, tension free mesh repair technique is regarded as gold standard. Based in the Stoppa technique, the laparoscopic hernia repair was developed in 1991. The most common laparoscopic techniques for inguinal hernia repair are transabdominal preperitoneal (TAPP) repair and total extraperitoneal (TEP) repair. The use of the laparoscopic technique was progressively increasing based on the advantages of minimal invasive procedures, but since the publication of Neumayer in 2004, where he reports a recurrent incidence in laparoscopic hernia of 10.1 % compared with 4% for open surgery, the use of laparoscopic repair declines considerably. Surgeons remain divided on the best technique for inguinal hernia repair: while more than half never perform laparoscopic inguinal hernia repair, today the laparoscopic technique for hernia repair is used in 28% of cases, of which 25% is used the TEP approach and is considered the best approach for bilateral inguinal hernia repair (17). Advantages and disadvantages of TEP are: faster return to usual activities, operation times are longer and there appears to be a higher risk of serious complication rate in respect of visceral (especially bladder) and vascular injuries (18).

In 1999, Gilbert published the use of bilayer patch device, known as prolene ® hernia system (Ethicon; Somerville, NJ, USA) (PHS) to repair inguinal hernia. The unique feature of this polypropylene mesh device is that it has attached the component, its underlay patch provides a pre-peritoneal repair, a connector that has the desirable attributes of a plug and an onlay patch covers the back wall. In the literature, better results have been reported for PHS repair than for Lichtenstein repair. The advantages of the anterior repair of inguinal hernias are: low operative costs, short learning curve, reproducible results at all levels and the possibility of the use of local anesthesia.

The objective of this study is to compare the results of laparoscopic totally extra-peritoneal repair (LTEPR) with open prolene hernia system repair (OPHSR) retrospectively.

DETAILED DESCRIPTION:
In our environment, 10367 (10.41% of all surgeries) hernia repair are performed in one year, of witch 5797 (51.92%) are inguinal hernia repair, of them 2870 (49.51%) are performed laparoscopically and 2927 (50.49%) are performed using different open repair techniques.

All consecutive patients that underwent LTEPR repair of inguinal hernia from 2003 to 2007 and open OPHSR inguinal hernia repair from 2008 to 2015, were analyzed. A total of 577 patients were included divided in two groups, the LTEPR group 293 patients and in the OPHSR group 284 patient. The selection of patients for LTEPR was bilateral inguinal hernia or recurrence after open repair, for OPHSR was unilateral inguinal hernia or health condition with preference to regional or local anesthesia. The follow up of all patients was between 18 to 60 months (mean 38.10 month).

Setting The LTEPR group was operated by two surgeons with long experience in laparoscopic hernia repair in a public hospital. The selected patients were those with bilateral inguinal hernia or recurrent hernia after open surgery, patients with contraindication for general anesthesia and patients with low midline scar or Pfannenstiel incision were excluded. Patients of the OPHSR group were operated in a private hospital by medical specialists in surgery with experience in repair using PHS; patients under local anesthesia were excluded.

Operative technique Pre-op antibiotic shot of 2rd generation cephalosporin was given to all the patients.

For LTEPR, under general anesthesia and supine position the plane preperitoneal was developed using a kidney-balloon trocar (Covidien-Medtronic, New Haven, CT, USA) using the 45 degrees scope to evaluate the plane. After developing the preperitoneal space, a structural trocar (Covidien-Medtronic, New Haven, CT, USA) was inserted and the space inflated with gas with low pressure. One working 10-millimeter trocar was inserted in the midline high as possible, if was necessary one more 5-millimeter trocar was inserted under the first one.

An atraumatic dissection of the groin was performed, the regional vessels (Corona Mortis, femoral and epigastric) were recognized, the cord was dissected and the peritoneal edge separated and retracted proximally wherever possible. A broad dissection was performed laterally including the Bogros space and superiorly releasing the peritoneum from the anterior abdominal wall.

To repair the groin, we use a heavyweight poli-propilene mesh 15X15 centimeters, divides in a piece of 15X5 centimeter inserted under the cord and fixed with helical tackers (Covidien-Medtronic, New Haven, CT, USA) to the ramus pubis and laterally to the transverse abdominal muscle. The second piece of mesh, 10X15 centimeter above the cord overlapping the anterior piece and fixing it to the rectus abdomini and to first mesh inserted. The gas was released and Bupivacaine Hydrochloride 0.5% was injected trough the trocar in the preperitoneal space.

For OPHSR, under regional or general anesthesia, in supine position, the groin was incised transversally, the planes were developed and after reduce de sac, the entry to the pre-peritoneal space was gained through the internal ring in indirect hernias, or medial defect in direct hernias. The preperitoneal space was the developed widely in atraumatic way. The posterior patch of the PHS was introduced pre-peritoneally and the onlay patch was fixed with continuous polypropylene sutures or separate stitches. Bupivacaine hydrochloride 0.5% was injected into the tissue around the repair.

This study was approved by the institution's ethics committee (Helsinki board). Statistical analysis All of the measured variables and derived parameters were tabulated using descriptive statistics. For the categorical variables, the summary tables provided the sample size, and absolute and relative frequencies. For the continuous variables, the summary tables provided the sample size, arithmetic mean, standard deviation, median, minimum and maximum values, and 95% confidence intervals (CI) for the means of the variables.

Analyses were performed using SPSS for Windows version 22.0 (SPSS, Chicago, IL, USA). Differences between two groups were analyzed using the Chi-square test, Fisher's exact test and t-test as adequate. Results were considered statistically significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* For laparoscopic repair: bilateral inguinal hernia or recurrent hernia For open repair: Patients with unilateral inguinal hernia More than 18 years old. Both sexes

Exclusion Criteria:

* Patient under 18 years old Patients who cannot sign the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent laparoscopic (TEP) repair with bilateral or recurrent hernia or open PHS repair with unilateral hernia or contraindication for general anesthesia .
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Pain scale | 60 months
  the patients were asked to classified their pair after surgery in visual analog scale from 0 to 10, being 0: no pain and 10 severe pain. (0: no pain, 1 to 3: mild pain, 4 to 6: moderate pain, and 7 to 10 severe pain.
complication after surgery | 60 months
  Complications were recorded from the records: type and number. Each type of complication is presented in a number of occurrences and calculates the percent of occurrence.

SECONDARY OUTCOMES:
Diary activity performance | 60 months
  patients were asked to respond about diary activity performing: no changes when the patient continues with the same job and sports activities improved: when the patient can do their normal activities without symptoms or sports activities, and worse: when the patients can not do their normal activities at all and are symptomatic.
Scar satisfaction | 60 months
  very satisfied- satisfied and unsatisfied depending in a subjective appreciation of the patients
sexual function | 60 months
  Better than before surgery, no changes or worse depending in can do their normal sexual function without symptoms, better or worse than before.

CONTACTS AND LOCATIONS:
Overall Officials: sergio Susmallian, MD, Principal Investigator — Assuta Medical Center
Locations (1):
- ASSUTAMC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
Data collected includes: names, type of surgery' complication, pain assessment, readmissions, satisfaction with the results, preoperative ASA clasification , postoperative hernia classification.
Time Frame: 60 months